CLINICAL TRIAL: NCT06436274
Title: Efficacy of Human Papillomavirus (HPV) Vaccination to Prevent Infection Among Women Living With HIV: A Prospective, Individual, Double-Blind, Randomized Controlled Study.
Brief Title: Efficacy of Human Papillomavirus (HPV) Vaccination to Prevent Infection Among Women Living With HIV.
Acronym: HOPE II
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Witwatersrand, South Africa (Other); Botswana Harvard Health Partnership (Unknown); Ministry of Health, Rwanda (Other Government); Fred Hutchinson Cancer Center (Other); National Cancer Institute (NCI) (NIH); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ruanne Barnabas, MBChB, MSc, DPhil., Chief of the Division of Infectious Diseases, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024P000880
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Human Papilloma Virus; Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into two different Groups. Group 1: Will receive nonavalent HPV vaccine at Day 0 and meningococcal vaccine at Month 18. Group 2: Will receive the meningococcal vaccine at Day 0 and nonavalent HPV at Month 18.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Will receive GARDASIL®9 vaccine at Day 0 and Menveo®/Menactra® vaccine at Month 18
  Interventions: Biological: GARDASIL®9; Biological: Menveo®/Menactra®
- Group 2 (Active Comparator): Will receive the Menveo®/Menactra® vaccine at Day 0 and GARDASIL®9 at Month 18
  Interventions: Biological: GARDASIL®9; Biological: Menveo®/Menactra®

INTERVENTIONS:
Biological: GARDASIL®9 — GARDASIL®9 or equivalent vaccines will be used for this study. These are FDA-approved vaccines.
Biological: Menveo®/Menactra® — Menveo®/Menactra® or equivalent vaccines will be used for this study. These are FDA-approved vaccines.

SUMMARY:
The Efficacy of Human Papillomavirus (HPV) Vaccination to Prevent Infection Among Women Living with HIV: A Prospective, Individual, Double-Blind, Randomized Controlled Study is evaluating immediate or delayed single-dose nonavalent HPV vaccination among women living with HIV who received prior HPV vaccination.

DETAILED DESCRIPTION:
The HOPE II Study is an individual-level, randomized trial of immediate or delayed vaccination with a single-dose of the nonavalent HPV vaccine. The primary outcome is single-dose HPV 16/18/31/33/45/52/58 vaccine efficacy (VE). The study will provide evidence on the efficacy of single-dose HPV 16/18/31/33/45/52/58 vaccination among women living with HIV.

Participants will be randomized 1:1 into two different Groups.

* Group 1: Will receive nonavalent HPV vaccine at Day 0 and meningococcal vaccine at Month 18
* Group 2: Will receive the meningococcal vaccine at Day 0 and nonavalent HPV at Month 18

The meningococcal vaccine was chosen as the control vaccination because meningococcal vaccination has no activity against HPV infection. Further, the meningococcal vaccine has the potential to be of benefit in a meningitis outbreak context and could be beneficial for young persons in a congregate setting such as tertiary institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16 years and above on the day of signing the ICF
2. Living with HIV with confirmed test results or clinic records
3. History of receiving HPV vaccine
4. Self-reported sexually active in the last six months
5. Lives within the study area and willing to provide updated locator information over the course of the study
6. Does not have an autoimmune, degenerative, or genetic disease
7. Does not have known advanced HIV (as per stage IV WHO clinical staging criteria for HIV)
8. No other Investigator-determined factor would limit participation in the trial
9. Has not and is not enrolled in a monoclonal, investigational vaccine, or a large quantity blood draw study
10. The participant has a cervix

Exclusion Criteria:

1. Anyone with cervical abnormality on examination
2. Anyone with an allergy to vaccine components or yeast

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Assigned female at birth
Enrollment: 778 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of single-dose HPV among women living with HIV who were vaccinated against HPV 16/18. | 18 Months
  Efficacy will be measured by the incidence of persistent infection from at least one of these HPV 16/18/31/33/45/52/58, where persistence is defined as a positive test at two consecutive visits at least 4.5 months apart.

SECONDARY OUTCOMES:
Safety and tolerability of single-dose nonavalent HPV vaccination in women living with HIV. | 18 Months
  This will be evaluated by comparing the occurrence of serious adverse events reported among each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Ruanne Barnabas, MBChB, MSc, DPhil, Principal Investigator — Massachusetts General Hospital; Sinead Delany-Moretlwe, MBBCh, PhD, DTM&H, Principal Investigator — Wits RHI, University of The Witwatersrand
Locations (3):
- Botswana Harvard Health Partnership, Gaborone, Botswana
- Ministry of Health and Center for Family Health Research, Kigali, Kigali, Rwanda
- Wits RHI, University of the Witwatersrand, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No